CLINICAL TRIAL: NCT03976193
Title: Improving Physical Activity Maintenance Following an Exercise Program for Cancer Survivors
Brief Title: Improving Physical Activity Maintenance of Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-0323.cc; P30CA046934 (NIH)
Record Dates: First submitted 2019-05-22; First posted 2019-06-05 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Cancer
Keywords: active treatment; Recent treatment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BfitBwell program (Placebo Comparator): BfitBwell is a 3-month supervised exercise program for cancer survivors delivered at the Anschutz Health and Wellness Center. This program has demonstrated effectiveness for improving physical fitness, fatigue, and depression among participants
  Interventions: Behavioral: BfitBwell program
- BfitBwell + 6, bi-weekly PA Behavior Change counseling session (Active Comparator): Participants randomized to BfitBwell + PA behavior change counseling sessions will receive six, 1-1.5 hour sessions lead by a Certified Exercise Physiologist, trained on the study protocol. Sessions will be held once per week, every other week at the Anschutz Health and Wellness center. Participants will attend the sessions in groups, as schedules allow. Behavior change discussion topics will target self-efficacy for exercise, barriers to exercise, goal setting, behavior modification strategies, time management, cognitive reframing, and relapse prevention. Participants in this study arm will receive a group education workbook in congruence to discussion session topics to promote notetaking, and self-reflective journaling.
  Interventions: Behavioral: BfitBwell program; Behavioral: 6 bi-weekly PA Behavior Change counseling sessions

INTERVENTIONS:
Behavioral: BfitBwell program — Well known behavior change strategies such as goal setting, and identifying barriers to PA can improve long term adherence to PA, and have been shown to enhance PA maintenance after completion of a supervised intervention among cancer survivors
Behavioral: 6 bi-weekly PA Behavior Change counseling sessions — Well known behavior change strategies such as goal setting, and identifying barriers to PA can improve long term adherence to PA, and have been shown to enhance PA maintenance after completion of a supervised intervention among cancer survivors
  Arms: BfitBwell + 6, bi-weekly PA Behavior Change counseling session

SUMMARY:
Participants enrolled in the BfitBwell Cancer Exercise Program at the University of Colorado Cancer Center will be randomized 1:1 to receive the current BfitBwell program, or BfitBwell plus six, group-based behavior change counseling sessions adapted from BEAT Cancer. We will stratify the randomization based on sex.

ELIGIBILITY:
Inclusion Criteria:

1. current patient at the University of Colorado Cancer Center
2. signed physician clearance to participate in a supervised exercise program
3. participant is actively receiving medical cancer treatment (chemotherapy, radiation or surgery) OR within 6 months of receiving medical cancer treatment.
4. Willingness to be randomized to receive six, PA behavior change counseling sessions as part of the BfitBwell program, and able to attend five out of six of these sessions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Examine the effects of six, group-based physical activity (PA) behavior change counseling sessions PA change from post-program, to 3-months following completion of the BfitBwell program. | 3 months
  The primary outcome will be self-reported weekly minutes of moderate to vigorous leisure-time PA, three-months following completion of the program, measured by the Godin Shepherd Leisure Time Exercise Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- UCD Anschutz Health and Wellness Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No